CLINICAL TRIAL: NCT00343512
Title: Pilot Study of Neoadjuvant Dose Dense Docetaxel With Correlative Molecular Studies in Stage II/III Breast Cancer
Brief Title: Docetaxel Followed by Surgery in Treating Women With Stage II or Stage III Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed due to competing neoadjuvant studies for a small patient population
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bapsi Chak, MD, Associate Professor; Radiation Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BRE 0368; VICC-BRE-0368; VICC-11239
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Results first posted 2010-11-09 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Docetaxel; Biopsy; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therapeutic Intervention (Experimental)
  Interventions: Drug: docetaxel; Genetic: protein expression analysis; Other: laboratory biomarker analysis; Procedure: biopsy; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: docetaxel — Docetaxel 75 mg/m2 IV (1-hour infusion) on day 1 of each cycle (cycle = 2 weeks) x 4 cycles
  Other Names: Taxotere
Genetic: protein expression analysis — protein expression analysis
Other: laboratory biomarker analysis — laboratory biomarker analysis
Procedure: biopsy — biopsy
Procedure: conventional surgery — conventional surgery
Procedure: neoadjuvant therapy — neoadjuvant therapy

SUMMARY:
RATIONALE: Dose-dense scheduling with (peg)filgrastim support may improve the clinical and pathologic complete response rate (pCR) and safety profile of single agent neoadjuvant docetaxel therapy.

PURPOSE: To evaluate whether dose-dense scheduling with (peg)filgrastim support may improve the clinical and pathologic complete response rate (pCR) and safety profile of single agent neoadjuvant docetaxel therapy. To determine the changes in molecular markers that occurs with single agent docetaxel, tissue will be obtained at the end of the four cycles of docetaxel (either by repeat biopsy or definitive surgery).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Pathologic complete response rate (pCR) of dose dense docetaxel in the neoadjuvant setting.

Secondary

* Safety and toxic effects of this regimen in these patients.
* Tumor response rate (as measured by ultrasound) in patients treated with this regimen.
* Determine whether early changes in markers of cell cycle position, proliferation, or apoptosis correlate with pathologic complete response rate in these patients.
* Determine whether the molecular profile that predicts for chemoresponsiveness also predicts for response to radiotherapy (as measured by local recurrence) in these patients.
* Determine whether tumors that demonstrate the greatest degree of change in protein expression patterns from pre- to post-docetaxel treatment will also be those that are most sensitive to chemotherapy (as measured by pathologic response rate) in these patients.

OUTLINE: This is a nonrandomized, open-label, pilot study.

* Tissue Collection: Patients undergo tumor core biopsy (6-8 cores) and blood collection prior to initiating neoadjuvant docetaxel.
* Neoadjuvant docetaxel with hematopoietic support: Patients receive docetaxel IV over 1 hour on day 1. Patients also receive pegfilgrastim subcutaneously (SC) on day 1 or 2 of each course OR filgrastim (G-CSF) or sargramostim (GM-CSF) SC daily beginning between day 2-4 of each course and continuing until blood counts recover. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Surgery: Within 4-6 weeks after completion of neoadjuvant docetaxel, patients undergo definitive surgery.

Patients undergo tumor biopsy and blood collection periodically for pharmacokinetic, genetic, and molecular biomarker correlative studies. Samples are examined for changes in p21 protein expression (and/or p21 phosphorylation) and the protein expression profile.

After completion of study treatment, patients are followed at least every 6 months for 3 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion:

* Histologically or cytologically confirmed invasive carcinoma of the breast by core biopsy
* Tumor ≥ 2 cm in greatest dimension(may be either node positive or node negative disease
* Patients with non-metastatic breast cancer who are in the judgment of the treating medical oncologist considered to be of sufficiently high risk to warrant adjuvant chemotherapy

  * Patients with internal mammary, supraclavicular and/or axillary node involvement are eligible. Patients with inflammatory breast cancer are eligible
  * Patients with T0 disease but palpable and measurable adenopathy are eligible for this trial. All sites of disease should be noted and followed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Menopausal status not specified
* Female ≥ 18 years old
* Absolute neutrophil count ≥ 1,000/mm^3
* Hemoglobin ≥ 8 g/dL
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin normal
* Alkaline phosphatase (AP), AST, and ALT meeting 1 of the following criteria:

  * AP normal AND AST or ALT ≤ 5 times ULN
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal
* Women of child-bearing potential, must have a negative serum pregnancy test and must use effective contraception for the duration of the study and for at least 6 months after completion of study treatment
* Patients with prior malignancies are eligible if they have been disease free for ≥ 5 years. Patients with curative treatment of non-melanomatous skin cancer, carcinoma in situ of the cervix, contralateral DCIS treated with mastectomy are eligible even if it is diagnosed in < 5 years.

PRIOR CONCURRENT THERAPY:

* No prior anthracycline or taxane-based chemotherapy. Patients who received chemoprevention are eligible if the chemopreventive agent has been discontinued for at least one year prior to enrollment in the current study.
* At least 1 year since prior tamoxifen for breast cancer prevention

Exclusion:

* Prior radiotherapy to the ipsilateral breast

  * Patients who have had radiation to the contralateral breast are eligible
* Evidence of distant metastatic disease (i.e., lung, liver, bone, brain)
* Pregnant of breastfeeding
* Patients who have congestive heart failure, angina pectoris, uncontrolled cardiac arrhythmia, or other significant heart disease, or who have had a myocardial infarction within the past year
* Patients with > grade 1 peripheral neuropathy
* Patients with a history of hypersensitivity reaction to products containing polysorbate 80 (Tween 80)
* Patients receiving an investigational anticancer drug within 3 weeks of registration
* Patients with serious medical illness that in the judgment of the treating physician, places the patient at risk.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-02; Primary Completion 2008-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from February 2004 to September 2007.
Pre-assignment Details: A total of 39 people were consented, one of which was ineligible. Four patients withdrew from the study before beginning treatment.
Groups:
- Therapeutic Intervention: Docetaxel 75 mg/m2 IV (1-hour infusion) on day 1 of each cycle (cycle = 2 weeks) x 4 cycles
Period: Overall Study
Arm/Group | Therapeutic Intervention
Started | 34
Completed | 32
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number Participants to Achieve Pathologic Complete Response
Description: whether or not patient has pathologic complete response (pCR) to dose dense docetaxel in the neoadjuvant setting (pCR = no residual viable tumor on histologic analysis)
Time Frame: 3 month
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 34
participants
  pCR: Yes | 5
  pCR: No | 29

2. Secondary Outcome: Safety Profile Based on Number of Patients With Each Worst-grade Toxicity
Description: Not all participants necessarily have an adverse event, thus not everyone will be accounted for in worst-grade toxicities. Likewise, one participant can potentially have more than one event in various grades 1-5 which accounts for the difference in number of patients analyzed and total number in the worst-grade toxicity tables. Tables represent the number of patients with worst-grade toxicity at each of five grades (grade 1, least severe; to grade 5, most severe) following NCI Common Toxicity Criteria
Time Frame: Through 30 days after completion of treatment
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 12
participants
  No. patients with worst-grade toxicity 1 | 5
  No. patients with worst-grade toxicity 2 | 8
  No. patients with worst-grade toxicity 3 | 11
  No. patients with worst-grade toxicity 4 | 1
  No. patients with worst-grade toxicity 5 | 0

3. Secondary Outcome: Tumor Response as Measured by Ultrasound
Description: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: At screening, 8 weeks and at surgery (within 14-21 days)
Measure: Number; unit: participants
Arm/Group | Therapeutic Intervention
Number analyzed (Participants) | 18
participants
  Complete Response | 5
  Progressive Disease | 1
  Stable Disease | 1
  Partial Response | 11

ADVERSE EVENTS:
Arm/Group | Therapeutic Intervention
Serious Adverse Events (participants affected / at risk) | 9/32
Other Adverse Events (participants affected / at risk) | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=32)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 1 (1)
Infection (Infections and infestations) | 6 (6) — possible port infections, dental infection
Vomiting (Gastrointestinal disorders) | 2 (2)
Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
pain, right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
hemoglobin increased (Investigations) | 6 (7)
fever (General disorders) | 2 (2)
edema, arm (General disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
hypertension (Vascular disorders) | 1 (2)
alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
bruising (Injury, poisoning and procedural complications) | 1 (2)
hypothyroidism (Endocrine disorders) | 1 (2)
nausea (Gastrointestinal disorders) | 2 (3)
hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
acute vascular leak syndrome (Vascular disorders) | 1 (1)
nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
alkaline phosphatase increase (Investigations) | 1 (1)
neuropathy (Nervous system disorders) | 2 (2)
sinus tachacardia (Cardiac disorders) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
weight loss (Investigations) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Intervention (N=32)
Allergic reaction (Immune system disorders) | 2 (7)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alkaline Phosphatase (Investigations) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (23)
ALT, SGPT (Metabolism and nutrition disorders) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
AST, SGOT (Metabolism and nutrition disorders) | 2 (2)
Blood, bone marrow (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Depression (Psychiatric disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry eye syndrome (Eye disorders) | 4 (4)
Dsypnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspepsia, heartburn (Gastrointestinal disorders) | 3 (3)
Edema (General disorders) | 4 (7)
Fatigue (General disorders) | 22 (25)
Flushes (Vascular disorders) | 8 (9)
Glucose, serum-high (Metabolism and nutrition disorders) | 7
Hemoglobin (Investigations) | 14 (15)
Hemorrhage (Vascular disorders) | 5 (5)
Infection (Infections and infestations) | 10 (11)
Insomnia (Psychiatric disorders) | 7 (7)
Irregular menses (Reproductive system and breast disorders) | 8 (8)
Leukocytes, (Blood and lymphatic system disorders) | 2 (2)
Memory impairment (Psychiatric disorders) | 3 (3)
Muscle weakness, legs (Musculoskeletal and connective tissue disorders) | 5 (8)
Musculoskelatal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 17 (17)
Nausea (Gastrointestinal disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 18 (25)
Pain - breast (General disorders) | 5 (5)
Pain, bone (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain, extermity limb (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain, headache (General disorders) | 4 (4)
Potassium, serum-low (Metabolism and nutrition disorders) | 4 (4)
Pruritus, itching (Skin and subcutaneous tissue disorders) | 2 (3)
Skin dry (Skin and subcutaneous tissue disorders) | 8 (9)
Skin reaction, hand-foot (Skin and subcutaneous tissue disorders) | 4 (6)
Sweating (General disorders) | 3 (3)
Taste alteration, dysgeusia (Nervous system disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 2 (2)
Watery eye, tearing (Eye disorders) | 10 (11)
Weight gain (Investigations) | 4 (4)
obesity (Metabolism and nutrition disorders) | 2 (2)
Weight loss (Investigations) | 3 (5)

LIMITATIONS AND CAVEATS:
All adverse events have been included in the "other adverse event" section. They are not differentiated by causality (eg. related to disease, con-meds).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes